CLINICAL TRIAL: NCT04996784
Title: Pharmacokinetics of Dexamethasone in COVID-19 Obese Patients
Acronym: CoDEX
Status: Completed | Type: Observational
Sponsor: Jules Desmeules (Other)
Responsible Party: Sponsor-Investigator, Jules Desmeules, Director, Head of Clinical pharmacology,Investigator, Clinical Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 2021-00034
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: Dexamethasone; Pharmacokinetics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal weight: The patients (n=30) will be stratified into 2 groups based on their body mass Index (BMI).The normal weight group will contain 15 patients with a 18.5 ≤ BMI ≤ 25 kg/m2.
  Each group will be divided in two subgroups (female/ male)
  Interventions: Other: Capillary blood sampling
- Obese: The patients (n=30) will be stratified into 2 groups based on their body mass Index (BMI). The obese group will contain 15 patients with a BMI ≥ 30 kg/m2.
  Each group will be divided in two subgroups (female/ male)
  Interventions: Other: Capillary blood sampling

INTERVENTIONS:
Other: Capillary blood sampling — The capillary blood sample will be obtained by pricking the fingertip using contact-activated lancet (BD Microtainer). A total of five blood drops (10 μL each) will be collected by a micropipette and will be dropped off on the blotting paper 903 S&S (Whatman).

SUMMARY:
In this regard, the present research project aims to compare dexamethasone PK in normal-weight versus obese patients treated for COVID-19.

This observational study will include patients hospitalized at HUG (Division of General Internal Medicine) with COVID-19 and treated with oral DEX. This study will include 2 groups of patients according to their body mass index (BMI) (normal weight with a BMI of 18.5-25.0 kg/m2; obese/ morbidly obese with a BMI ≥30). The primary outcome will be the assessment of the differential impact of weight on DEX PK. Finally, the data generated will be used to build a physiologically based PK (PBPK) model for DEX and in different sub-groups. The model will aim to predict the effect of BMI in virtual populations with different drugs and in different scenarios. This should allow prospective dose adjustment of DEX based on patient weight.

DETAILED DESCRIPTION:
Before starting the study, COVID-19 patients receiving dexamethasone as part of their hospital management and meeting the criteria of inclusion and non-exclusion will have an information session with an investigator as described above.

During the study session, capillary blood samples will be taken during a total of 8 hours, time starting just before DEX administration, and at the following times after the dose: time of the drug intake, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours and 8 hours. The capillary blood sample will be obtained by pricking the fingertip using contact-activated lancet (BD Microtainer). A total of five blood drops (10 μL each) will be collected by a micropipette and will be dropped off on the blotting paper 903 S&S (Whatman). After a 45-minute drying time at room temperature, dried blood samples (DBS) samples will be packed in sealable plastic bags containing a desiccant and stored at - 80°C until analysis. Drugs will be extracted from DBS using methanol. DEX quantification in capillary DBS will be performed using reverse-phase- HPLC coupled to tandem mass spectrometer (MS/MS). In addition to this, an EDTA tube (3 ml) of blood will be collected and preserved in the biobank (-80°C) and will be used whether further analysis should be performed on the samples. In this aim an authorization to reuse the samples will be requested from each patient during the consent signature.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years receiving DEX for COVID-19
* Stable dose of DEX for at least 24 hours
* BMI between 18.5 and 25 or ≥ 30 kg/m2
* Understanding of French orEnglish languages and ability to give a written inform consent

Exclusion Criteria:

* Medical history of cirrhosis (Child Pugh B and C) or/and nonalcoholic fatty liver disease.
* History of bariatric or other gastric surgery that may affect the drug absorption
* Patient already included in a clinical trial of an investigational drug
* Use of drugs that may affect CYP3A activity * *based on the 'drug interactions and cytochromes P450' table published by The Division of clinical Pharmacology and Toxicology [15], HUG and on the investigator's knowledge and on the drug interactions website from the University of Liverpool (https://www.covid19- druginteractions.org/checker).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty COVID-19 hospitalized patients will be informed and included in the study after giving a written informed consent. The control group will include mainly normal weight patients (BMI 18.5- 25 kg/m2) receiving DEX.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
AUC comparison | 8 hours
  The primary endpoint will be the AUC of DEX determined after a 6 mg oral dose at steady state.

SECONDARY OUTCOMES:
PK parameters | 8 hours
  Extrapolation from the AUC values of the Dexamethasone Clearance in the two groups
PK parameters | 8 hours
  Extrapolation from the AUC values of the Dexamethasone Cmax in the two groups
PK parameters | 8 hours
  Extrapolation from the AUC values of the Dexamethasone T1/2 in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- University hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No